CLINICAL TRIAL: NCT03488628
Title: High-Flow Nasal Oxygen Therapy for Exacerbation of Chronic Pulmonary Obstructive Disease: A Randomized, Open-label, Single-center, Pilot Study.
Brief Title: High-Flow Nasal Oxygen Therapy for Exacerbation of Chronic Pulmonary Obstructive Disease.
Acronym: OxyCOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2017-16; ID RCB: 2017-A03535-48 (Other: French Ministry of Health)
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: respiratory failure; oxygen therapy; Noninvasive ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noninvasive ventilation (Active Comparator): Noninvasive ventilation delivered through a face mask, in alternance with standard nasal oxygen therapy
  Interventions: Other: Noninvasive ventilation
- High-Flow Nasal Oxygen therapy (Experimental): High-Flow Nasal Oxygen therapy delivered continuously over the first 24 hours by the AIRVO2® device (Fisher & Paykel Healthcare,New Zealand) through nasal canula.
  Interventions: Other: High-Flow Nasal Oxygen therapy

INTERVENTIONS:
Other: Noninvasive ventilation — Noninvasive ventilation delivered through a face mask, in alternace with satandard nasal oxygen therapy over the first 24 hours
  Arms: Noninvasive ventilation
Other: High-Flow Nasal Oxygen therapy — High-Flow Nasal Oxygen therapy delivered continuously over the first 24 hours by the AIRVO2® device (Fisher & Paykel Healthcare,New Zealand) through nasal canula.
  Arms: High-Flow Nasal Oxygen therapy

SUMMARY:
High-Flow Nasal Oxygen (HFNO) therapy has never been tested against Noninvasive ventilation, the reference standard therapy for acute exacerbation of chronic obstructive pulmonary disease (COPD), in randomized clinical trials.

The aim of the present study is to compare the effects of HFNO therapy on arterial blood gas variables over the first 24 hours of therapy, to those of Noninvasive ventilation, in patients experiencing a moderate (i.e. with arterial pH within 7.25-7.35) exacerbation of COPD.

DETAILED DESCRIPTION:
As soon as admission to the intensive care unit, eligible patients who gave consent will be randomized to either HFNO or Noninvasive ventilation therapy for at least the first 24 hours.

In the usual care group , Noninvasive ventilation will be applied in alternance with standard nasal oxygen therapy.

In the intervention group, HFNO with be applied continuously over the first 24 hours.

In both groups, an oxygen saturation, as assessed by finger pulse oximetry, of 88-92% will be targeted.

The primary objective will be two-fold: to compare between groups 1) Efficacy, assessed by the arterial pH at 24 hours, and 2) Safety, assessed by the ratio of the arterial partial pressure in oxygen (PaO2) over the inspired oxygen fraction (FiO2) at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Known Chronic Obstructive Pulmonary disease (COPD)
* respiratory rate or presence of accessory respiratory muscles activity on physical exam
* moderate exacerbation of COPD as defined by an arteria pH between 7.25 and 7.35 and an arterial carbon dioxide partial pressure (PaCO2) equal or above 45 mm Hg

Exclusion Criteria:

* Age below 18
* Pregnancy
* Known sleep apnea syndrome
* Patent treated by noninvasive ventilation at home
* Not affiliated to French scial security
* Contraindication to aither Noninvasive ventilation or to High-Flow Nasal Oxygen therapy
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Arterial pH at 24 hours | 24 hours
  Arterial pH at 24 hours, the primary efficacy criteria, is planned to be jointly assessed and analysed with the primary safety criteria (PaO2/FiO2 ratio at 24 hours)
PaO2/FiO2 ratio at 24 hours | 24 hours
  PaO2/FiO2 ratio at 24 hours, the primary safety criteria, is planned to be jointly assessed and analysed with the primary efficacy criteria (arterial pH at 24 hours)

SECONDARY OUTCOMES:
Cumulative incidence of tracheal intubation | 28 days
  Cumulative incidence of tracheal intubation from randomisation through Day 28, with discharge alive or death (without having been intubated) before day 28 handled as competing events
Time course of arterial pH | 24 hours
  Arterial pH will be measured 5 times over the first 24 hours (before application of the randomized intervention, 1 hour after and then at H6, H12 and H24)
Arterial partial pressure in carbon dioxide (PaCO2) | 24 hours
  PaCO2 be measured 5 times over the first 24 hours (before application of the randomized intervention, 1 hour after and then at H6, H12 and H24)
Time course of arterial oxygen saturation (SaO2) | 24 hours
  SaO2 will be measured by oximetry on arterial blood samples, 5 times over the first 24 hours (before application of the randomized intervention, 1 hour after and then at H6, H12 and H24)
Self-reported dyspnea score | 24 hours
  Patients will grade their dyspnea every 6 hours on a 5-point numeric scale (ranging from -2 [marked worsening] to +2 [frank improvement])
Perceived nursing workload | 24 hours
  Nurses will rate perceived workload on a 100 mm-visual numeric scale (ranging from 0 [negligible workload] to 100 mm [the most demanding task ever experienced] every 4 hours
Proportion of patients who will need Noninvasive ventilation in the High-Flow Nasal Oxygen group from randomisation through the 24th hour | 24 hours
  Need of Noninvasive ventilation in the High-Flow Nasal Oxygen group
Severe Adverse events | 28 days
  Severe Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh Nay, MD, Principal Investigator — Centre Hospitalier Régional d'Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No